CLINICAL TRIAL: NCT03865953
Title: A Phase IIa Study of the Efficacy and Safety of Oral LAT8881 in Neuropathic Pain
Brief Title: Oral LAT8881 in Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lateral Pharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAT-NP-001; 2018-004534-15 (EudraCT Number)
Record Dates: First submitted 2019-03-02; First posted 2019-03-07 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-04

CONDITIONS: Neuropathic Pain; Diabetic Peripheral Neuropathy (DPN); Post Herpetic Neuralgia (PHN)
MeSH Terms: conditions — Neuralgia; Neuralgia, Postherpetic

STUDY DESIGN:
Intervention Model Description: This is the first study with LAT8881 in subjects with neuropathic pain. As such, it has been designed to evaluate, in a well-defined patient group, the concept that LAT8881 is safe and effective in this indication.
  Subjects enrolled into this study have been diagnosed with Post Herpetic Neuralgia (PHN) or Diabetic Peripheral Neuropathy (DPN), both conditions being well accepted examples of neuropathic pain. Because the pain is chronic, without a period effect, and treatment is symptomatic rather than curative, a crossover study is considered appropriate. Studies with other agents have successfully demonstrated analgesic effects in PHN and DPN with a crossover study design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LAT8881 (Active Comparator): 1 x 30 mg capsule of LAT8881 taken by mouth, twice daily (morning and evening) during the four-week treatment period.
  Interventions: Drug: LAT8881
- Placebo (Placebo Comparator): 1 x 30 mg capsule of placebo, taken by mouth, twice daily (morning and evening) during the four-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LAT8881 — LAT8881 oral capsule
  Arms: LAT8881
Drug: Placebo — Placebo oral capsule
  Arms: Placebo

SUMMARY:
This is a randomised, placebo-controlled, double-blind, crossover, phase IIa study to investigate the efficacy and safety of oral LAT8881 in neuropathic pain.

DETAILED DESCRIPTION:
This is a randomised, placebo-controlled, double-blind, crossover, phase IIa study to investigate the efficacy and safety of oral LAT8881 in neuropathic pain. After a one week baseline period, subjects entered into the study will be randomised to receive Investigational Medicinal Product (IMP) (LAT8881 or placebo) twice daily for four weeks.

The first treatment period will be followed by a washout period of two weeks and then a second baseline period of one week. Subjects will not take any IMP over these three weeks.

After the second baseline period, subjects will cross over to receive the second treatment (either LAT8881 or placebo, whichever treatment was not received in the first treatment period) twice daily for four weeks.

The pharmacokinetics (PK) of LAT8881 will be investigated in 15 subjects (PK subjects) at selected Australian sites.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of post herpetic neuralgia, with pain persisting for at least 3 months after the onset of herpes zoster rash OR
2. Clinical diagnosis of distal painful polyneuropathy due to Type I or Type II diabetes mellitus with:

   1. symmetrical, bilateral pain in the lower extremities for at least 3 months and
   2. diabetes under control for at least 3 months prior to randomisation, as indicated by a glycated haemoglobin level (HbA1c) of ≤ 11% (97 mmol/mol) and on a stable dose of insulin or oral diabetic medication for 3 months prior to screening, and
   3. no change in diabetic medication planned for the duration of the study
3. Positive sensory symptoms (mechanical or thermal) associated with neuropathic pain, confirmed by:

   1. painDETECT questionnaire (PD-Q) and
   2. Clinical assessment, showing signs of neuropathic pain in either a dermatomal (PHN) or distal symmetrical distribution (DPN)

8. An average daily pain score on the numeric pain rating scale (NPRS) of at least 4 and no more than 8 in the last five diary entries before randomisation

Exclusion Criteria:

1. Presence of moderate to severe pain from other causes that may confound assessment or self-evaluation of NP.
2. Subjects with both DPN and PHN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (4):
  - Paratus Clinical Research Kanwal, Kanwal, New South Wales
  - Paratus Clinical Research Blacktown, Sydney, New South Wales
  - AusTrials, Brisbane, Queensland
  - Emeritus Research Services, Melbourne, Victoria
- United Kingdom (2):
  - University of Bristol, Bristol
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No
This is an Early Proof of Concept study

RESULTS

PARTICIPANT FLOW:
Groups:
- LAT8881, Then Placebo: In the first intervention period, 1 x 30 mg capsule of LAT8881 was taken twice daily (morning and evening) for four weeks. After a 3 week washout/baseline non-treatment period, a placebo capsule was taken twice daily (morning and evening) for four weeks.
- Placebo, Then LAT8881: In the first intervention period, a placebo capsule was taken twice daily (morning and evening) for four weeks. After a 3 week washout/baseline non-treatment period, 1 x 30 mg capsule of LAT8881 was taken twice daily (morning and evening) for four weeks.
Period: First Intervention (4 Weeks)
Arm/Group | LAT8881, Then Placebo | Placebo, Then LAT8881
Started | 25 | 28
Completed | 23 | 27
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 0 | 1
Period: Washout/Baseline Period (3 Weeks)
Arm/Group | LAT8881, Then Placebo | Placebo, Then LAT8881
Started | 23 | 27
Completed | 23 | 27
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | LAT8881, Then Placebo | Placebo, Then LAT8881
Started | 23 | 27
Completed | 23 | 25
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAT8881, Then Placebo | Placebo, Then LAT8881 | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.33) | 58.5 (8.91) | 59.8 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 10 | 21 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 12
  Australia | 19 | 22 | 41
Neuropathic pain history [Count of Participants; unit: Participants]
  Post herpetic neuralgia (PHN) | 8 | 2 | 10
  Diabetic peripheral neuropathy (DPN) | 17 | 26 | 43
PainDETECT questionnaire (PD-Q) scores [Mean (Standard Deviation); unit: units on a scale] — The painDETECT questionnaire (PD-Q) is used to assist in identifying patients with neuropathic pain. It consists of seven pain sensory symptom items which are scored from 0 "not at all" to 5 "very strongly" plus one pain course pattern item scored from -1 to 2 and and one pain radiation item scored as 2 or 0. From this questionnaire, a PD-Q total score, ranging from -1 to 38 is calculated. A total score ≥19 indicates a neuropathic component is likely, ≤12 indicates a neuropathic component is unlikely and scores 13-18 are considered uncertain.
  units on a scale | 21.0 (3.62) | 20.9 (5.03) | 20.9 (4.38)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Pain Score, Using an 11 Point Numeric Pain Rating Scale (NPRS)
Description: The 11-point numeric pain rating scale (NPRS) ranges from 0 ("no pain") to 10 ("worst pain imaginable"). A larger negative number represents a greater reduction in pain.
  The efficacy of oral LAT8881 in neuropathic pain was compared with placebo, when assessed by change in mean pain intensity scores, using this 11 point numeric pain rating scale.
Time Frame: Baseline to Week 4
Population: The per protocol population was used for all efficacy analyses. This population excluded subjects with inadequate exposure to treatment or who had other major protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale | -0.87 (1.53) | -0.74 (2.09)
Statistical Analysis 1: Comparison: LAT8881 vs Placebo; Subject numbers gave a 90% power to demonstrate a statistically significant difference in the mean change from baseline NPRS for the active treatment compared with placebo of at least 1 unit, with a two sided test at a 5% level of significance; Test type: Superiority — Analysis used a two-period two-treatment crossover design; p = 0.67, Mixed Models Analysis; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.76 to 0.49]

2. Secondary Outcome: Change in NPRS Score After the First and Last Dose of LAT8881 and Placebo
Description: To investigate the effect of oral LAT8881 in neuropathic pain compared with placebo, as measured by the numeric pain rating score (NPRS). The 11-point numeric pain rating scale ranges from 0 ("no pain") to 10 ("worst pain imaginable"). A larger negative number represents a greater reduction in pain.
  This outcome was investigated only in the pharmacokinetic subset of per protocol subjects.
Time Frame: Pre-dose, 0.5,1,2,4 and 6 hours after the first and last dose of LAT8881 and placebo
Population: Pharmacokinetic subset of the per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 14 | 14
score on a scale
  Absolute baseline score, first dose | 4.5 (2.2) | 4.8 (1.9)
  Change from baseline, 0.5 hours after first dose | -0.1 (0.77) | -0.2 (1.53)
  Change from baseline, 1 hour after first dose | -0.4 (0.63) | -0.6 (1.95)
  Change from baseline, 2 hours after first dose | -0.1 (0.95) | -0.8 (2.26)
  Change from baseline, 4 hours after first dose | 0.1 (1.07) | -0.6 (2.17)
  Change from baseline, 6 hours after first dose | 0.0 (0.68) | -0.7 (1.77)
  Absolute baseline score, last dosing day | 4.4 (2.2) | 4.0 (2.2)
  Change from baseline, 0.5 hours after last dose | -0.6 (2.43) | -0.4 (0.84)
  Change from baseline, 1 hour after last dose | -0.5 (2.58) | -0.4 (1.02)
  Change from baseline, 2 hours after last dose | -0.8 (2.19) | -0.1 (0.77)
  Change from baseline, 4 hours after last dose | -0.5 (2.26) | -0.4 (0.93)
  Change from baseline, 6 hours after last dose | -0.7 (1.93) | -0.4 (0.84)

3. Secondary Outcome: Change in Mean Pain Scores After 1, 2 and 3 Weeks of Treatment, Using NPRS
Description: To investigate the effect of oral LAT8881 on mean pain scores in neuropathic pain compared with placebo, as measured by the numeric pain rating scale (NPRS). The 11-point numeric pain rating scale ranges from 0 ("no pain") to 10 ("worst pain imaginable"). A larger negative number represents a greater reduction in pain.
Time Frame: 1,2 and 3 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
units on a scale
  Baseline | 6.18 (1.53) | 6.18 (1.45)
  Change from baseline at Week 1 | -0.50 (1.37) | -0.55 (1.27)
  Change from baseline at Week 2 | -0.73 (1.49) | -0.91 (1.62)
  Change from baseline at Week 3 | -0.84 (1.61) | -0.84 (1.88)

4. Secondary Outcome: 30% Responder Rate in Oral LAT8881 Compared With Placebo, as Assessed by the Numeric Pain Rating Scale.
Description: To determine the proportion of subjects with at least a 30% reduction in mean NPRS after 4 weeks treatment. The 11-point numeric pain rating scale (NPRS) ranges from 0 ("no pain") to 10 ("worst pain imaginable"). A decrease in pain score represents an improvement in pain.
Time Frame: 4 weeks
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
Participants | 20 | 19

5. Secondary Outcome: 50% Responder Rate in Oral LAT8881 Compared With Placebo, as Assessed by the Numeric Pain Rating Scale.
Description: To determine the proportion of subjects with at least a 50% reduction in mean the numeric pain rating scale (NPRS) after 4 weeks treatment. The 11-point numeric pain rating scale ranges from 0 ("no pain") to 10 ("worst pain imaginable"). A decrease in pain score represents an improvement in pain.
Time Frame: 4 weeks
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
Participants | 6 | 9

6. Secondary Outcome: Maximum Change in Mean NPRS
Description: To determine the maximum effects of oral LAT8881 in neuropathic pain, compared with placebo, as measured by the numeric pain rating scale (NPRS). The 11-point numeric pain rating scale ranges from 0 ("no pain") to 10 ("worst pain imaginable"). A larger negative number represents a greater reduction in pain..
Time Frame: 1,2,3 or 4 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale | -1.53 (1.37) | -1.55 (1.41)

7. Secondary Outcome: Change in Functioning as Assessed by the Brief Pain Inventory Interference Scale (BPI)
Description: To evaluate the effects of oral LAT8881, compared with placebo, on functioning when measured by the Brief Pain Inventory Interference Scale (BPI). The BPI assesses the severity of pain and its impact on functioning. Patients are asked to assess the level of interference experienced across seven items; general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life, with a "0" meaning "no interference, and a "10", at the top end of the scale, meaning "complete interference". The result is the mean of the score of the seven items. A reduction in mean score indicates a decrease in interference.
Time Frame: 4 weeks
Population: Per protocol population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline BPI | 4.71 (2.45) | 4.91 (2.32)
  Change from baseline | -0.57 (1.83) | -1.12 (1.97)

8. Secondary Outcome: Change in Pain Characteristics and Intensity, as Assessed by the Short Form McGill Pain Questionnaire (SF-MPQ-2)
Description: To evaluate the effect of oral LAT8881, compared with placebo, on pain symptoms in subjects with neuropathic pain, when measured by the Short Form McGill Pain Questionnaire (SF-MPQ-2). The SF-MPQ-2 contains 22 descriptors of pain and related symptoms, each scored from "0" (none) to "10" (worst possible). The scores for each descriptor at each visit are averaged to give a mean score from 0 to 10. A larger negative number represents a greater reduction in pain.
Time Frame: 4 weeks
Population: Per protocol population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline SF-MPQ-2 | 3.88 (1.81) | 3.86 (1.73)
  Change from baseline | -0.66 (1.34) | -0.63 (1.70)

9. Secondary Outcome: Change in Neuropathic Pain Symptoms, as Assessed by Neuropathic Pain Symptom Inventory (NPSI)
Description: The Neuropathic Pain Symptom Inventory (NPSI) contains ten items related to different pain descriptors (e.g. burning, squeezing, electric-shock, stabbing, tingling), allowing the assessment of the different dimensions of neuropathic pain, and two items related to the frequency and duration of pain. Each pain descriptor is rated on an 11-point numeric rating scale from 0 (no pain) to 10 (worst imaginable pain). Total pain intensity score is calculated by the sum of the 10 descriptors and can range from 0 to 100. A higher score indicates a higher pain intensity. A larger negative number represents a greater reduction in pain.
Time Frame: 4 weeks
Population: Per protocol population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline NPSI | 40.7 (17.2) | 41.1 (16.2)
  Change from baseline | -6.0 (14.5) | -7.4 (16.9)

10. Secondary Outcome: Change in Emotional Functioning, as Assessed by the Beck Depression Inventory-II
Description: To evaluate the effect of oral LAT8881, compared with placebo, on emotional functioning when measured by the Beck Depression Inventory-II (BDI-II). The BDI-II consists of 21 items; each item is a list of four statements arranged in order of increasing severity about a particular symptom of depression. Each statement is scored from 0 to 3. Each of the 21 items is summed to give a single score for the BDI-II. Scores can range from 0 (no depression) to 63 (severe depression). An increase from baseline to the end of treatment indicates a deterioration.
Time Frame: 4 weeks
Population: Per protocol population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  Baseline BDI-II | 11.3 (8.6) | 12.1 (9.3)
  Change from baseline | -1.1 (4.14) | -1.2 (7.98)

11. Secondary Outcome: Patient Global Impression of Change Score
Description: The Patient Global Impression of Change (PGIC) is a a single-item rating by subjects of their improvement with treatment during a clinical trial. It asks the subject to rate their improvement with therapy on a 7-point scale, ranging from substantially worse ("0") to substantially improved ("7"), with no change ("4") as the mid-point. A score above 4 indicates an improvement.
Time Frame: 4 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale | 4.5 (1.23) | 4.8 (1.33)

12. Secondary Outcome: Rescue Medication Use
Description: To determine the change from baseline in paracetamol rescue medication use during oral LAT8881 administration, compared with placebo.
Time Frame: Weekly over four-week treatment
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 53 | 53
gram
  Week 1 | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline. | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline.
  Week 2 | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline. | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline.
  Week 3 | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline. | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline.
  Week 4 | NA (NA) — Only one subject took additional paracetamol rescue medication (1 g/day on three days only). Due to this limited use of rescue medication, it was not considered appropriate to calculate rescue medication use per week for the group compared with baseline. | NA (NA) — No subjects took additional paracetamol rescue medication, compared with baseline.

13. Secondary Outcome: Maximum Plasma Concentration of LAT8881 (Cmax) After Oral LAT8881
Description: Cmax is calculated after the first dose of IMP on Day 1 and after 4 weeks treatment on the morning of Day 28
Time Frame: Day 1 and Day 28
Population: Subgroup of the pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 3 | 3
ng/mL
  Cmax, Day 1 | NA (NA) — Cmax could not be calculated as the majority of samples were below the limit of quantification. | NA (NA) — Cmax could not be calculated as the majority of samples were below the limit of quantification.
  Cmax, Day 28 | NA (NA) — Cmax could not be calculated as the majority of samples were below the limit of quantification. | NA (NA) — Cmax could not be calculated as the majority of samples were below the limit of quantification.

14. Secondary Outcome: Time to Maximum Plasma Concentration of LAT8881 (Tmax)
Description: Tmax after the first dose of investigational medicinal product (IMP) and after 4 weeks treatment with IMP
Time Frame: Day 1 and day 28
Population: subgroup of the pharmacokinetic population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 3 | 3
hours
  Tmax, Day 1 | NA (NA) — Tmax could not be calculated as the majority of samples were below the limit of quantification. | NA (NA) — Tmax could not be calculated as the majority of samples were below the limit of quantification.
  Tmax, Day 28 | NA (NA) — Tmax could not be calculated as the majority of samples were below the limit of quantification. | NA (NA) — Tmax could not be calculated as the majority of samples were below the limit of quantification.

15. Secondary Outcome: Area Under the Concentration Time Curve From Zero to Infinity (AUC0-inf)
Description: AUC0-inf after the first dose of IMP and after 4 weeks of treatment
Time Frame: Day 1 and Day 28
Population: Subgroup of the pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 3 | 3
ng-hr/mL
  AUC0-inf, Day 1 | NA (NA) — AUC0-inf could not be calculated as the majority of samples were below the limit of quantification. | NA (NA) — AUC0-inf could not be calculated as the majority of samples were below the limit of quantification.
  AUC0-inf, Day 28 | NA (NA) — AUC0-inf could not be calculated as the majority of samples were below the limit of quantification. | NA (NA) — AUC0-inf could not be calculated as the majority of samples were below the limit of quantification.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study treatment until the End of Study visit, maximum 93 days
Arm/Group | LAT8881 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 5/51 | 6/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAT8881 (N=51) | Placebo (N=51)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for legal reasons, the investigator will not reveal the result of the study to a third party without a mutual agreement about the analysis and interpretation of the data with the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT03865953/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03865953/SAP_001.pdf